CLINICAL TRIAL: NCT05437172
Title: Clinical and Radiographic Evaluation of Autogenous Demineralized Dentin Graft for Ridge Preservation With and Without Injectable Platelet Rich Fibrin (A Randomized Controlled Clinical Trial)
Brief Title: Evaluation of Autogenous Demineralized Dentin Graft for Ridge Preservation With and Without Injectable Platelet Rich Fibrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Odai Amer Ahmad Hwafdeh, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Shaam
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Ridge Preservation; Alveolar Bone Loss; Dentin Graft
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- injectable platelet rich fibrin with deminerlized dentin graft (Experimental): injectable platelet rich fibrin with deminerlized dentin graft for ridge preservation after teeth extraction
  Interventions: Procedure: injectable platelet rich fibrin with demineralized dentin graft
- deminerlized dentin graft (Active Comparator): deminerlized dentin graft for ridge preservation after teeth extraction
  Interventions: Procedure: demineralized dentin graft

INTERVENTIONS:
Procedure: injectable platelet rich fibrin with demineralized dentin graft — after atraumatic extraction, collection of whole venous blood (9 ml) in sterile vacutainer tubes will be done without anticoagulant added, vacutainer tubes will be then placed in a centrifugal machine at 700 revolutions per minute (rpm) for 3 min with a tube filled with water to maintain the balance during the centrifuging process. ADDG particles prepared by demineralization of tooth particles in 0.6N hydrochloric acid for 30 min to achieve demineralization then washed twice in saline and dried with sterile gauze. Graft particles will be loaded at the defect site to restore ridge form, large metal condenser was used to adapt the graft to the defect and stabilizing the graft with sutures.
  Arms: injectable platelet rich fibrin with deminerlized dentin graft
Procedure: demineralized dentin graft — after atraumatic extraction, ADDG particles will be prepared by demineralization of tooth particles in 0.6N hydrochloric acid for 30 min to achieve demineralization then washed twice in saline and dried with sterile gauze.
  Graft particles will be loaded at the defect site to restore ridge form, large metal condenser was used to adapt the graft to the defect and stabilizing the graft with sutures.
  Arms: deminerlized dentin graft

SUMMARY:
Ridge preservation should be considered whenever possible after tooth extraction. Whether implant placement would be performed or for aesthetic consideration at pontic sites when conventional bridge is planned. Ridge preservation aims to maximize the bone formation accompanied with good soft tissue architecture to facilitate implant and prosthetic replacement restoring function, phonetics and aesthetics. the Aim of the study is To evaluate the bucco-lingual ridge width clinically and radiographically, height of buccal and lingual ridges of the socket after application of injectable platelet rich fibrin and autogenous dentin graft.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years need of at least one single rooted tooth extraction.
* Non-restorable teeth.
* Systemically healthy patients.
* Good oral hygiene, Plaque index less than 15%.
* Non-smoker or Smoking ≤ 10 cigarettes/day.
* Cooperative patients able and accept to come for follow up appointments.

Exclusion Criteria:

* Any interim intervention that may have affected any of the outcomes of interest.
* Pregnant and lactation females.
* Smoking ˃ 10 cigarettes/day.
* Patients reporting systemic conditions that may compromise healing or bone metabolism (eg: diabetes).
* Patients with poor oral hygiene.
* Any known allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Radiographic Bucco-lingual ridge width change | up to 24 weeks
  radiographic measurement

SECONDARY OUTCOMES:
Changes in the height of the socket buccal and lingual ridges. | up to 24 weeks
  radiographic measurement
postoperative pain | immediately after the procedure
  Visual analogue scale from zero (better) to 10 (worse)
Patient satisfaction | immediately after the procedure
  binary yes and no
Keratinized tissue width | up to 24 weeks
  periodontal probe measurement
chair time | immediately after the procedure
  in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Odai A Hwafdeh, BDS, Principal Investigator — Master student; Nesma M Shemais, PhD, Study Director — Lecturer of Oral Medicine and Periodontology, Faculty of Dentistry, Cairo University; Mona S Darhous, PhD, Study Chair — Professor of Oral Medicine and Periodontology, Faculty of Dentistry, Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Manial, Egypt

IPD SHARING:
Plan to Share IPD: Undecided